CLINICAL TRIAL: NCT00113386
Title: Phase III Randomized Trial of Preoperative Chemotherapy Versus Preoperative Concurrent Chemotherapy and Thoracic Radiotherapy Followed by Surgical Resection and Consolidation Chemotherapy in Favorable Prognosis Patients With Stage IIIA (N2) Non-Small Cell Lung Cancer
Brief Title: Cisplatin and Docetaxel With or Without Radiation Therapy in Treating Patients Who Are Undergoing Surgery for Newly Diagnosed Stage III Non-Small Cell Lung Cancer
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: This study terminated early due to low accrual.
Sponsor: Radiation Therapy Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH); SWOG Cancer Research Network (Network); Cancer and Leukemia Group B (Network); Eastern Cooperative Oncology Group (Network); North Central Cancer Treatment Group (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RTOG-0412; CDR0000429479; SWOG-S0332; CALGB-RTOG-0412; ECOG-RTOG-0412; NCCTG-RTOG-0412
Record Dates: First submitted 2005-06-07; First posted 2005-06-08 (Estimated); Results first posted 2012-12-27 (Estimated); Last update posted 2013-06-28 (Estimated); Status verified 2013-06

CONDITIONS: Lung Cancer
Keywords: stage IIIA non-small cell lung cancer; adenocarcinoma of the lung; large cell lung cancer; squamous cell lung cancer; bronchoalveolar cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Adenocarcinoma of Lung; Adenocarcinoma, Bronchiolo-Alveolar | interventions — Filgrastim; pegfilgrastim; Cisplatin; Docetaxel; Chemotherapy, Adjuvant; Neoadjuvant Therapy; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Induction chemotherapy, surgery, consolidation chemotherapy (Other): Induction/surgery/consolidation
  Interventions: Biological: filgrastim; Biological: pegfilgrastim; Drug: cisplatin; Drug: docetaxel; Procedure: adjuvant therapy; Procedure: conventional surgery; Procedure: neoadjuvant therapy
- Chemotherapy and radiation, surgery, consolidation ch (Other): Induction/radiation/surgery/cosolidation
  Interventions: Biological: filgrastim; Biological: pegfilgrastim; Drug: cisplatin; Drug: docetaxel; Procedure: adjuvant therapy; Procedure: conventional surgery; Procedure: neoadjuvant therapy; Radiation: radiation therapy

INTERVENTIONS:
Biological: filgrastim — Consolidation chemotherapy
Biological: pegfilgrastim — Consolidation chemotherapy
Drug: cisplatin
Drug: docetaxel
Procedure: adjuvant therapy
Procedure: conventional surgery
Procedure: neoadjuvant therapy
Radiation: radiation therapy
  Arms: Chemotherapy and radiation, surgery, consolidation ch

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as cisplatin and docetaxel, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Radiation therapy uses high-energy x-rays to kill tumor cells. Cisplatin and docetaxel may make tumor cells more sensitive to radiation therapy. Giving more than one drug (combination chemotherapy) together with radiation therapy before surgery may shrink the tumor so it can be removed. Giving chemotherapy after surgery may kill any tumor cells that remain after surgery. It is not yet known whether giving cisplatin and docetaxel together with radiation therapy is more effective than giving cisplatin together with docetaxel in treating non-small cell lung cancer.

PURPOSE: This randomized phase III trial is studying cisplatin, docetaxel, and radiation therapy to see how well they work compared to cisplatin and docetaxel in treating patients who are undergoing surgery for newly diagnosed stage III non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare overall survival of patients with newly diagnosed favorable prognosis stage IIIA non-small cell lung cancer treated with neoadjuvant cisplatin and docetaxel with vs without thoracic conformal radiotherapy followed by surgical resection and docetaxel.

Secondary

* Compare median and progression-free survival of patients treated with these regimens.
* Compare clinical and pathologic response rates in patients treated with these regimens.
* Compare the toxicity of these regimens in these patients.
* Correlate pathological complete response with disease-free and overall survival of patients treated with these regimens.
* Correlate DNA damage repair genes (ERCC1 and XRCC1), microtubule-related proteins (TUBB-III and MAP4), and shed tumor DNA with response and outcome in patients treated with these regimens.
* Correlate protein profiles, using MALDI-TOF proteomic analysis of tumor and serum, with response and prognosis in patients treated with these regimens.
* Compare quality of life of patients treated with these regimens.
* Determine the efficacy of fludeoxyglucose F 18 positron emission tomography scanning in assessing pathological response of the tumor and the mediastinal lymph nodes and in predicting long-term outcome in patients treated with these regimens.
* Correlate comorbid conditions with survival of patients treated with these regimens.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to T stage (T1 vs T2-3), number of involved mediastinal lymph nodes (1 vs 2 or more vs not evaluable), and nodal micrometastases vs clinically involved nodes (mN2 vs cN2).

* Induction therapy: Patients are randomized to 1 of 2 treatment arms.

  * Arm I: Patients receive cisplatin IV over 1 hour and docetaxel IV over 1 hour on days 1 and 22.
  * Arm II: Patients undergo thoracic conformal radiotherapy once daily 5 days a week for approximately 5½ weeks (total of 28 doses). Patients also receive cisplatin IV over 1 hour on days 1, 8, 22, and 29 and docetaxel IV over 1 hour on days 1, 8, 15, 22, and 29.
* Surgery: Within 4-8 weeks after completion of induction therapy, patients with stable disease or better undergo a lobectomy or pneumonectomy with a formal systematic mediastinal lymph node dissection.
* Consolidation therapy: Beginning 4-6 weeks after surgery, patients receive docetaxel IV over 1 hour on days 1, 22, and 43 and pegfilgrastim or filgrastim (G-CSF) subcutaneously on days 2, 23, and 44.

Quality of life is assessed at baseline, within 2 weeks after completion of induction therapy, and then at 6 and 12 months after surgery.

After completion of study treatment, patients are followed every 3 months for 1 year, every 6 months for 2 years, and then annually thereafter.

PROJECTED ACCRUAL: A total of 574 patients will be accrued for this study within 4 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed primary non-small cell lung cancer (NSCLC)*, including any of the following cellular types:

  * Adenocarcinoma
  * Squamous cell carcinoma
  * Large cell carcinoma
  * Non-lobar and non-diffuse bronchoalveolar cell carcinoma
  * NSCLC not otherwise specified NOTE: *Diagnosed within the past 3 months; diagnosis by mediastinal nodal biopsy or needle aspiration allowed provided a distinct lung primary (separate from the nodes) is clearly evident on CT scan
* Stage IIIA disease

  * T1-T3 disease

    * If pleural effusion is present, must meet ≥ 1 of the following criteria to exclude T4 disease:

      * Pleural effusion cytologically negative by thoracentesis
      * Documented absence of pleural metastases and pleural effusion cytologically negative by thoracoscopy (for patients with pleural effusion on CT scan [but not on chest x-ray] that is deemed too small to tap safely under either CT scan or ultrasound guidance)
  * Confirmed positive ipsilateral mediastinal lymph node(s) (N2 disease)**, with or without positive ipsilateral hilar nodes, by mediastinoscopy, mediastinotomy, endoscopic ultrasound-guided transesophageal biopsy, thoracotomy, video-assisted thoracoscopy, Wang needles, or fine needle aspiration under bronchoscopic or CT guidance

    * N2 nodes must be separate from primary tumor by CT scan or surgical exploration AND maximum diameter ≤ 3.0 cm
    * Mediastinoscopy OR other means of mediastinal lymph node biopsy required (regardless of the primary tumor site) for patients with subcarinal lymphadenopathy by size criteria or by positron emission tomography (PET) scan
    * If the lymph nodes in the contralateral mediastinum and neck are visible by contrast CT scan of the chest AND are ≥ 1.0 cm OR if contralateral involvement is suggested by PET scan, lymph nodes must be confirmed negative by one of the above diagnostic procedures AND N3 status must be confirmed negative by histology or cytology
    * No palpable lymph nodes in the supraclavicular areas or higher in the neck unless proven benign by excisional biopsy
    * A nodal biopsy or needle aspiration may be omitted provided all of the following criteria are true:

      * Paralyzed left true vocal cord by bronchoscopy or indirect laryngoscopy
      * Nodes visible in the aortopulmonary window (level 5) region on CT scan
      * Distinct primary tumor (separate from the nodes) is visible by CT scan
      * No evidence of subcarinal nodal involvement by CT scan NOTE: **PET scan positivity is not sufficient to establish N2 nodal status
* Measurable disease by chest x-ray and/or contrast-enhanced CT scan
* Candidate for surgery

  * Resectable disease
* No distant metastases, including other ipsilateral or contralateral parenchymal lesions or liver or adrenal metastases, by history or physical examination, fludeoxyglucose F 18 PET scan, MRI or CT scan of the brain, chest x-ray and/or CT scan of the lungs and upper abdomen

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* Zubrod 0-1

Life expectancy

* Not specified

Hematopoietic

* Absolute neutrophil count ≥ 1,800/mm^3
* Platelet count ≥ 100,000/mm^3
* Hemoglobin ≥ 10.0 g/dL (transfusion or other intervention allowed)

Hepatic

* ALT and AST ≤ 2.5 times upper limit of normal (ULN)
* Alkaline phosphatase ≤ 2.5 times ULN
* Bilirubin ≤ 1.5 times ULN
* No hepatic insufficiency resulting in clinical jaundice or coagulation defects

Renal

* Creatinine clearance ≥ 60 mL/min

Cardiovascular

* No unstable angina or congestive heart failure requiring hospitalization within the past 6 months
* No transmural myocardial infarction within the past 6 months

Pulmonary

* FEV_1 ≥ 2.0 L OR
* Predicted post-resection FEV_1 ≥ 0.8 L
* DLCO ≥ 50% of predicted
* No chronic obstructive pulmonary disease exacerbation
* No other respiratory illness requiring hospitalization or that would preclude study therapy

Immunologic

* No AIDS
* No prior allergic reaction to the study drugs
* No history of severe hypersensitivity to other drugs formulated with polysorbate 80
* No acute bacterial or fungal infection requiring IV antibiotics

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No unintentional weight loss > 5% of body weight within the past 6 months
* No pre-existing peripheral neuropathy ≥ grade 2
* No other invasive malignancy within the past 3 years except nonmelanoma skin cancer or carcinoma in situ of the breast, oral cavity, or cervix
* No other severe active comorbidity

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No prior biological agent for this cancer
* No concurrent filgrastim (G-CSF), sargramostim (GM-CSF), or pegfilgrastim during study induction therapy (for patients randomized to the chemoradiotherapy arm)

Chemotherapy

* No prior systemic chemotherapy for this cancer

  * Prior chemotherapy for a different cancer allowed

Endocrine therapy

* Not specified

Radiotherapy

* No prior radiotherapy to the region of this cancer that would result in overlap of radiotherapy fields
* No routine post-operative radiotherapy
* No concurrent intensity modulated radiotherapy

Surgery

* See Disease Characteristics

Other

* No prior gefitinib for this cancer
* No concurrent amifostine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2005-04; Primary Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maria Werner-Wasik, MD, Principal Investigator — Sidney Kimmel Cancer Center at Thomas Jefferson University; Howard L. West, MD, Principal Investigator — Swedish Cancer Institute at Swedish Medical Center - First Hill Campus; Jeffrey Crawford, MD, Study Chair — Duke Cancer Institute; Chandra P. Belani, MD, Study Chair — University of Pittsburgh; James R. Jett, MD, Study Chair — Mayo Clinic
Locations (76):
- United States (76):
  - Cancer Center at Providence Alaska Medical Center, Anchorage, Alaska
  - Arkansas Cancer Research Center at University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Cancer Care Center at John Muir Health - Concord Campus, Concord, California
  - Moores UCSD Cancer Center, La Jolla, California
  - USC/Norris Comprehensive Cancer Center and Hospital, Los Angeles, California
  - University of California Davis Cancer Center, Sacramento, California
  - Memorial Hospital, Colorado Springs, Colorado
  - Front Range Cancer Specialists, Fort Collins, Colorado
  - Poudre Valley Hospital, Fort Collins, Colorado
  - CCOP - Christiana Care Health Services, Newark, Delaware
  - Mayo Clinic - Jacksonville, Jacksonville, Florida
  - Ella Milbank Foshay Cancer Center at Jupiter Medical Center, Jupiter, Florida
  - Watson Clinic, LLC, Lakeland, Florida
  - CCOP - Mount Sinai Medical Center, Miami Beach, Florida
  - Phoebe Cancer Center at Phoebe Putney Memorial Hospital, Albany, Georgia
  - CCOP - Atlanta Regional, Atlanta, Georgia
  - Northeast Georgia Medical Center, Gainesville, Georgia
  - Delnor Community Hospital - Geneva, Geneva, Illinois
  - Cardinal Bernardin Cancer Center at Loyola University Medical Center, Maywood, Illinois
  - Community Cancer Center, Normal, Illinois
  - Advocate Christ Medical Center, Oak Lawn, Illinois
  - Cancer Treatment Center at Pekin Hospital, Pekin, Illinois
  - Oncology Hematology Associates of Central Illinois, PC - Peoria, Peoria, Illinois
  - OSF St. Francis Medical Center, Peoria, Illinois
  - Cancer Institute at St. John's Hospital, Springfield, Illinois
  - Reid Hospital & Health Care Services, Incorporated, Richmond, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Hematology Oncology Associates of the Quad Cities, Bettendorf, Iowa
  - Genesis Regional Cancer Center at Genesis Medical Center, Davenport, Iowa
  - Markey Cancer Center at University of Kentucky Chandler Medical Center, Lexington, Kentucky
  - St. Agnes Hospital Cancer Center, Baltimore, Maryland
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Frederick Memorial Hospital Regional Cancer Therapy Center, Frederick, Maryland
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - CCOP - Michigan Cancer Research Consortium, Ann Arbor, Michigan
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - Upper Michigan Cancer Center at Marquette General Hospital, Marquette, Michigan
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - St. John's Regional Medical Center, Joplin, Missouri
  - St. John's Regional Health Center, Springfield, Missouri
  - Siteman Cancer Center at Barnes-Jewish Hospital, St Louis, Missouri
  - Good Samaritan Cancer Center at Good Samaritan Hospital, Kearney, Nebraska
  - Methodist Cancer Center at Methodist Hospital - Omaha, Omaha, Nebraska
  - UNMC Eppley Cancer Center at the University of Nebraska Medical Center, Omaha, Nebraska
  - Valley Hospital - Ridgewood, Ridgewood, New Jersey
  - NYU Cancer Institute at New York University Medical Center, New York, New York
  - SUNY Upstate Medical University Hospital, Syracuse, New York
  - Faxton Regional Cancer Center, Utica, New York
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - Leo W. Jenkins Cancer Center at ECU Medical School, Greenville, North Carolina
  - Lenoir Memorial Cancer Center, Kinston, North Carolina
  - FirstHealth Moore Regional Community Hospital Comprehensive Cancer Center, Pinehurst, North Carolina
  - Charles M. Barrett Cancer Center at University Hospital, Cincinnati, Ohio
  - Arthur G. James Cancer Hospital and Solove Research Institute at Ohio State University, Columbus, Ohio
  - Veterans Affairs Medical Center - Portland, Portland, Oregon
  - Oregon Health & Science University Cancer Institute, Portland, Oregon
  - St. Luke's Hospital Cancer Center, Bethlehem, Pennsylvania
  - Penn State Cancer Institute at Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Lancaster General Hospital, Lancaster, Pennsylvania
  - Kimmel Cancer Center at Thomas Jefferson University - Philadelphia, Philadelphia, Pennsylvania
  - Albert Einstein Cancer Center, Philadelphia, Pennsylvania
  - Allegheny Cancer Center at Allegheny General Hospital, Pittsburgh, Pennsylvania
  - York Cancer Center at Apple Hill Medical Center, York, Pennsylvania
  - Hollings Cancer Center at Medical University of South Carolina, Charleston, South Carolina
  - CCOP - Greenville, Greenville, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - U.T. Cancer Institute at University of Tennessee Medical Center, Knoxville, Tennessee
  - Medical City Dallas Hospital, Dallas, Texas
  - Simmons Comprehensive Cancer Center at University of Texas Southwestern Medical Center - Dallas, Dallas, Texas
  - CCOP - Virginia Mason Research Center, Seattle, Washington
  - Swedish Cancer Institute at Swedish Medical Center - First Hill Campus, Seattle, Washington
  - Madigan Army Medical Center - Tacoma, Tacoma, Washington
  - Vince Lombardi Cancer Clinic - Green Bay at Aurora BayCare Medical Center, Green Bay, Wisconsin
  - Dean Medical Center - Madison, Madison, Wisconsin
  - Vince Lombardi Cancer Clinic - Sheboygan, Sheboygan, Wisconsin

RESULTS

PARTICIPANT FLOW:
Groups:
- Preoperative Cisplatin/Docetaxel: Preoperative (induction) cisplatin/docetaxel; surgical resection 4-8 weeks post-chemotherapy; docetaxel 4-6 weeks post-surgery
- Preoperative Radiotherapy and Cisplatin/Docetaxel: Preoperative (induction) throacic radiation therapy 50.4 Gy concurrently with cisplatin/docetaxel; surgical resection 4-8 weeks post-chemotherapy and radiation therapy; docetaxel 4-6 weeks post-surgery.
Period: Overall Study
Arm/Group | Preoperative Cisplatin/Docetaxel | Preoperative Radiotherapy and Cisplatin/Docetaxel
Started | 10 | 9
Completed | 3 | 5
Not Completed | 7 | 4
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Physician Decision | 0 | 1
Not completed — Toxicity | 3 | 0
Not completed — Ineligible | 1 | 2
Not completed — Unknown - Lost to Follow-Up | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Preoperative Cisplatin/Docetaxel: Preoperative cisplatin/docetaxel; surgical resection 4-8 weeks post-chemotherapy; docetaxel 4-6 weeks post-surgery [Data is reported for eligible patients with on-study information, which is 8 patients.]
- Preoperative Radiotherapy and Cisplatin/Docetaxel: Preoperative throacic radiation therapy 50.4 Gy concurrently with cisplatin/docetaxel; surgical resection 4-8 weeks post-chemotherapy and radiation therapy; docetaxel 4-6 weeks post-surgery. [Data is reported for eligible patients with on-study information, which is 7 patients.]
- Total: Total of all reporting groups
Arm/Group | Preoperative Cisplatin/Docetaxel | Preoperative Radiotherapy and Cisplatin/Docetaxel | Total
Number analyzed (Participants) | 8 | 7 | 15
Age Continuous [Median (Full Range); unit: years] | 66 [43 to 77] | 57 [45 to 72] | 63 [43 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 | 6
  Male | 6 | 3 | 9

OUTCOME MEASURES:

1. Primary Outcome: Comparison of Overall Survival
Time Frame: Date of death or date of last follow-up
Population: This study terminated early with 19 out of 574 subjects accrued. Therefore no analysis was performed.
Groups:
- Preoperative Cisplatin/Docetaxel: Preoperative cisplatin/docetaxel; surgical resection 4-8 weeks post-chemotherapy; docetaxel 4-6 weeks post-surgery
- Preoperative Radiotherapy and Cisplatin/Docetaxel: Preoperative throacic radiation therapy 50.4 Gy concurrently with cisplatin/docetaxel; surgical resection 4-8 weeks post-chemotherapy and radiation therapy; docetaxel 4-6 weeks post-surgery.
Arm/Group | Preoperative Cisplatin/Docetaxel | Preoperative Radiotherapy and Cisplatin/Docetaxel
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Description: If a subject experienced more than one of a given SAE, the subject is counted only once for that SAE. If a subject experienced more than one of a given "Other (Not Includind Serious)" AE, then the subject is counted only once for that "Other (Not Including Serious)" AE.
Groups:
- Preoperative Cisplatin/Docetaxel: Preoperative cisplatin/docetaxel; surgical resection 4-8 weeks post-chemotherapy; docetaxel 4-6 weeks post-surgery. [Data is reported for eligible patients with adverse event information, which is 9 patients.]
- Preoperative Radiotherapy and Cisplatin/Docetaxel: Preoperative throacic radiation therapy 50.4 Gy concurrently with cisplatin/docetaxel; surgical resection 4-8 weeks post-chemotherapy and radiation therapy; docetaxel 4-6 weeks post-surgery. [Data is reported for eligible patients with adverse event information, which is 7 patients.]
Arm/Group | Preoperative Cisplatin/Docetaxel | Preoperative Radiotherapy and Cisplatin/Docetaxel
Serious Adverse Events (participants affected / at risk) | 5/9 | 4/7
Other Adverse Events (participants affected / at risk) | 7/9 | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Preoperative Cisplatin/Docetaxel (N=9) | Preoperative Radiotherapy and Cisplatin/Docetaxel (N=7)
Febrile neutropenia (Blood and lymphatic system disorders) | 4 | 0
Atrial flutter (Cardiac disorders) | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 1 | 0
Colonic hemorrhage (Gastrointestinal disorders) | 0 | 1
Rectal hemorrhage (Gastrointestinal disorders) | 0 | 1
Wound infection (Infections and infestations) | 1 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 1
Neutrophil count decreased (Investigations) | 4 | 1
Platelet count decreased (Investigations) | 1 | 0
White blood cell decreased (Investigations) | 3 | 0
Bronchial fistula (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary fistula (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypertension (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 1 | 1
Thromboembolic event (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Preoperative Cisplatin/Docetaxel (N=9) | Preoperative Radiotherapy and Cisplatin/Docetaxel (N=7)
Anemia (Blood and lymphatic system disorders) | 6 | 4
Blood and lymphatic system disorders - Other (Blood and lymphatic system disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0
Paroxysmal atrial tachycardia (Cardiac disorders) | 0 | 1
Sinus tachycardia (Cardiac disorders) | 0 | 2
Ventricular arrhythmia (Cardiac disorders) | 1 | 1
Ear and labyrinth disorders - Other (Ear and labyrinth disorders) | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 1 | 0
Flashing lights (Eye disorders) | 0 | 1
Retinal detachment (Eye disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 3
Diarrhea (Gastrointestinal disorders) | 5 | 1
Dyspepsia (Gastrointestinal disorders) | 1 | 1
Dysphagia (Gastrointestinal disorders) | 1 | 3
Esophagitis (Gastrointestinal disorders) | 0 | 4
Mucositis oral (Gastrointestinal disorders) | 2 | 0
Nausea (Gastrointestinal disorders) | 5 | 6
Oral pain (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 2 | 4
Chills (General disorders) | 1 | 0
Edema limbs (General disorders) | 1 | 1
Fatigue (General disorders) | 6 | 6
Fever (General disorders) | 2 | 1
Non-cardiac chest pain (General disorders) | 2 | 3
Pain (General disorders) | 0 | 1
Allergic reaction (Immune system disorders) | 1 | 0
Enterocolitis infectious (Infections and infestations) | 1 | 0
Infections and infestations - Other (Infections and infestations) | 2 | 0
Wound infection (Infections and infestations) | 1 | 0
Burn (Injury, poisoning and procedural complications) | 0 | 1
Dermatitis radiation (Injury, poisoning and procedural complications) | 0 | 1
Activated partial thromboplastin time prolonged (Investigations) | 1 | 0
Alanine aminotransferase increased (Investigations) | 1 | 1
Alkaline phosphatase increased (Investigations) | 1 | 2
Aspartate aminotransferase increased (Investigations) | 4 | 1
Creatinine increased (Investigations) | 2 | 1
Forced expiratory volume decreased (Investigations) | 0 | 1
Haptoglobin decreased (Investigations) | 2 | 0
INR increased (Investigations) | 1 | 0
Lymphocyte count decreased (Investigations) | 2 | 0
Neutrophil count decreased (Investigations) | 2 | 0
Platelet count decreased (Investigations) | 4 | 3
Weight loss (Investigations) | 1 | 2
White blood cell decreased (Investigations) | 4 | 2
Alkalosis (Metabolism and nutrition disorders) | 0 | 1
Anorexia (Metabolism and nutrition disorders) | 3 | 5
Dehydration (Metabolism and nutrition disorders) | 2 | 2
Hypercalcemia (Metabolism and nutrition disorders) | 0 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 3 | 3
Hyperkalemia (Metabolism and nutrition disorders) | 1 | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 | 1
Hypocalcemia (Metabolism and nutrition disorders) | 3 | 2
Hypokalemia (Metabolism and nutrition disorders) | 2 | 3
Hypomagnesemia (Metabolism and nutrition disorders) | 1 | 2
Hyponatremia (Metabolism and nutrition disorders) | 4 | 4
Hypophosphatemia (Metabolism and nutrition disorders) | 1 | 0
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Dizziness (Nervous system disorders) | 2 | 1
Dysgeusia (Nervous system disorders) | 0 | 2
Nervous system disorders - Other (Nervous system disorders) | 0 | 1
Peripheral motor neuropathy (Nervous system disorders) | 1 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 2
Agitation (Psychiatric disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 1
Confusion (Psychiatric disorders) | 0 | 1
Depression (Psychiatric disorders) | 2 | 0
Insomnia (Psychiatric disorders) | 2 | 2
Cystitis noninfective (Renal and urinary disorders) | 0 | 1
Urinary retention (Renal and urinary disorders) | 1 | 1
Erectile dysfunction (Reproductive system and breast disorders) | 0 | 1
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 3
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 | 4
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pharyngeal fistula (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 | 2
"Respiratory, thoracic and mediastinal disorders - Other" (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Alopecia (Skin and subcutaneous tissue disorders) | 2 | 2
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 2
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0
Purpura (Skin and subcutaneous tissue disorders) | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 1
Hypertension (Vascular disorders) | 1 | 1
Hypotension (Vascular disorders) | 1 | 1

LIMITATIONS AND CAVEATS:
This study terminated early with 19 out of 574 subjects accrued. Therefore no analysis was performed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No